CLINICAL TRIAL: NCT04129073
Title: QUO VADIS - QUality Of Life and surviVAl in carDIac arreSt Patients
Brief Title: QUality Of Life and surviVAl in carDIac arreSt Patients
Acronym: QUOVADIS
Status: Not yet recruiting | Type: Observational
Sponsor: Gruppo Italiano per la Valutazione degli Interventi in Terapia Intensiva (Other)
Responsible Party: Sponsor
Other Study IDs: QUO VADIS
Record Dates: First submitted 2019-10-11; First posted 2019-10-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Cardiac Arrest; Post-Anoxic Coma; Central Nervous System Diseases
Keywords: Comparative Effectiveness Research
MeSH Terms: conditions — Heart Arrest; Central Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac arrest patients admitted to Intensive Care treatment: Intensive Care treatment; Utilization of neuroprognostication tools
  Interventions: Other: Intensive care treatment

INTERVENTIONS:
Other: Intensive care treatment — Intensive care treatment; Utilization of neuroprognostication tools

SUMMARY:
QUO VADIS is a national observational study with the aim to describe clinical intervention and utilization of neuroprognostication tools in the management of patients admitted to ICU following cardiac arrest

DETAILED DESCRIPTION:
Despite recent improvements in post-resuscitation care, about 50% of patients resuscitated from cardiac arrest die or have poor neurological prognosis. Post-anoxic brain injury is common after cardiac arrest and is a major cause of post-resuscitation mortality. Since there has been a significant investment in improving the emergency response to both in-hospital ad out-of-hospital cardiac arrest (IHCA and OHCA, respectevly) patients and reported improvements in short-term survival outcomes, the long-term neurological state and quality of life of survivors and their caregiver is of growing significance.

QUO VADIS is a national observational study created to describe clinical interventions and utilization of neuroprognostication tools in the management of patients admitted to ICU following cardiac arrest.

The aims of the study are:

* To create an Italian Registry that describes clinical interventions and neuroprognostication tools used in the management of patients admitted to ICU following cardiac arrest
* To evaluate, after one year from the cardiac arrest, the neurological outcome and the quality of life of the patients;
* To evaluate, after one year from the cardiac arrest, the quality of life of caregivers;
* To identify the most effective clinical intervention in the management of post-cardiac arrest patients admitted to ICU;
* To create a prognostic model for patients admitted to ICU after cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 14 years;
* Cardiac Arrest within 24 hours ICU admission

Exclusion Criteria:

* Absence of Informed consent;
* Age < 14 years

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cardiac arrest patients admitted to ICU for specific care
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Disability | 6 months
  GOSe (Glascow Outcome Scale extended). Minimum value: 1 = Dead; Maximum value: 8= Upper Good Recovery
Neurological Outcome | 6 months
  mRS (modified Ranking Scale) Minimum value: 0 = Complete recovery; Maximum value: 6 = Death
Patients quality of life | 12 months
  EuroQoL-5D (european quality of life 5 dimensions). 0 = Worst imaginable health state; 100 = best imaginable health state

SECONDARY OUTCOMES:
Caregiver quality of life | 12 months
  Caregiver Burden Inventory. 0 to 20 = little or no burden; 61 to 88 = severe burden

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Livigni, MD, Principal Investigator — Ospedale San Giovanni Bosco, Turin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GiViTI website — http://www.giviti.marionegri.it/